CLINICAL TRIAL: NCT02553603
Title: The Effect of Growth Hormone Releasing Hormone on Cognitive Function in Individuals With Mild Cognitive Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-0086
Record Dates: First submitted 2015-09-03; First posted 2015-09-17 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Growth Hormone-Releasing Hormone; tesamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mild Cognitive Impairment, Placebo (Placebo Comparator): Subjects aged 55 - 85 years, scored between 23- 26 on screening Mini Mental Status Exam, receiving placebo Growth Hormone Releasing Hormone (GHRH).
  Interventions: Drug: Placebo Growth Hormone Releasing Hormone
- Non-cognitively impaired, Placebo (Placebo Comparator): Subjects aged 55- 85 years, scored between 27-30 on screening Mini Mental Status Exam, receiving placebo Growth Hormone Releasing Hormone (GHRH).
  Interventions: Drug: Placebo Growth Hormone Releasing Hormone
- Mild Cognitive Impairment, GHRH (Experimental): Subjects aged 55 - 85 years, scored between 23- 26 on screening Mini Mental Status Exam, receiving active Growth Hormone Releasing Hormone (GHRH).
  Interventions: Drug: Growth Hormone Releasing Hormone (GHRH)
- Non-cognitively impaired, GHRH (Experimental): Subjects aged 55 - 85 years, scored between 27-30 on screening Mini Mental Status Exam, receiving active Growth Hormone Releasing Hormone (GHRH).
  Interventions: Drug: Growth Hormone Releasing Hormone (GHRH)

INTERVENTIONS:
Drug: Growth Hormone Releasing Hormone (GHRH) — Growth Hormone Releasing Hormone (GHRH) 1mg/day for 10 weeks
  Other Names: Egrifta; tesamorelin
  Arms: Mild Cognitive Impairment, GHRH; Non-cognitively impaired, GHRH
Drug: Placebo Growth Hormone Releasing Hormone — Placebo GHRH to be given once daily for 10 weeks
  Other Names: Placebo
  Arms: Mild Cognitive Impairment, Placebo; Non-cognitively impaired, Placebo

SUMMARY:
This study is examining the effects of growth hormone releasing hormone (GHRH) on mild cognitive impairment (MCI). GHRH will be given at a dose of 1mg/day for 10 weeks to subjects with MCI as well as healthy controls.

DETAILED DESCRIPTION:
Subjects with MCI as well as healthy controls will be given GHRH at a dose of 1mg/day for 10 weeks.

This study is designed to investigate the effects of GHRH on the following things: 1) cognitive function as measured by our neuropsychologist with a series of short tests; 2) brain activity as measured by fMRI 3) lean and fat mass of your body as measured by DEXA; 4) physical function as measured by a walking test.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 to ≤ 85 years
* Ability to sign consent form (score ≥ on the Mini Mental State Examination, MMSE)
* MCI group: MMSE scores of 23 - 26
* Normal Control Group: MMSE scores of 27 - 30

Exclusion Criteria:

* Diabetes
* A neurologic condition other than MCI which might cause cognitive impairment
* Baseline serum IGF-1 concentration greater than the midrange for healthy young adults (300ng/ml)
* Presence of a pacemaker or metal implant
* Heart Failure
* Edema
* Active malignancy
* Carpal tunnel syndrome
* Disruption of the hypothalamic pituitary axis such that the pituitary is expected to be insensitive to growth hormone secretagogues such as GHRH
* Known allergy to tesamorelin or mannitol
* Pregnancy
* Significant heart, liver, kidney, blood or respiratory disease
* Active cancer
* Recent (within 6 months) treatment with anabolic steroids, GHRH or corticosteroids
* Alcohol or drug abuse
* MMSE < 23
* Less than 12 years of education
* Significant findings on screening tests, including but not limited to, blood counts, blood biochemistries, urinalysis, drug screening, HIV test, hepatitis panel, electrocardiogram
* Other medical conditions deemed exclusionary by the study investigators

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Cognitive Function measured by SLUMS | 10 weeks
  Cognitive function at 10 weeks measured by the St Louis University Mental Status (SLUMS)
Brain Perfusion measured by fMRI | 10 weeks
  Brain Perfusion at 10 week measured by MRI
Brain Morphology measured by MRI | 10 weeks
  Brain Morphology at 10 weeks measured by MRI

SECONDARY OUTCOMES:
Body composition measured by DEXA | 10 weeks
  Body composition at 10 weeks measured by DEXA
Physical Function measured by 6 minute walking test | 10 weeks
  Physical Function at 10 weeks measured by 6 minute walking test

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Urban, MD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States